CLINICAL TRIAL: NCT00181259
Title: In Vivo Cardiac Metabolism in Normal, Ischemic, and Cardiomyopathic Patients During Rest and Stress
Brief Title: Magnetic Resonance Spectroscopy Studies of Cardiac Muscle Metabolism
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00044690; R01HL061912-14 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure, Congestive
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The metabolism of the heart provides the chemical energy needed to fuel ongoing normal heart contraction. Magnetic resonance spectroscopy is a technique used in a MRI scanner that can be used to measure and study heart metabolism directly but without blood sampling or obtaining tissue biopsies. One of the hypotheses this study aims to investigate is whether energy metabolism is reduced in heart failure and whether that contributes to the poor heart function.

DETAILED DESCRIPTION:
This study uses magnetic resonance (MR) spectroscopy to study heart metabolism and function in normal subjects and patients with left ventricular hypertrophy, dilated cardiomyopathy, and those with coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Healthy subjects: no history of heart disease
* Dilated cardiomyopathy: history of heart failure, ejection fraction (EF) <40%
* Left ventricular hypertrophy: wall thickness >1.2cm
* Coronary artery disease: >50% coronary lesion or positive stress test

Exclusion Criteria:

* contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease, dilated cardiomyopathy, or left ventricular hypertrophy
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1988-01; Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Phosphocreatine/adenosine triphosphate (PCr/ATP) and creatine kinase (CK) flux | At time of magnetic resonance spectroscopy (MRS)
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?

SECONDARY OUTCOMES:
Phosphocreatine (PCr) | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
ATP | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
[Cr] or total creatine (CR), or CR/water ratio | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
Sodium (NA) | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
ATP flux | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
31P distribution or metabolite map | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
23Na distribution or metabolite map | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?
CR distribution or metabolite map | At time of MRS
  Can non-invasive magnetic resonance imaging and spectroscopy techniques be developed, validated, and implemented on clinical MR scanners in order to address the questions of a.) the extent to which myocardial high-energy phosphate (HEP), creatine (Cr), or sodium concentrations change in response to and after transient ischemia or chronic ischemic injury, b.) the extent to which myocardial high-energy phosphates, creatine, or sodium concentrations as well as HEP flux are altered in cardiomyopathic patients with and without/ congestive heart failure, c.) can spatial differences in cardiac metabolites (HEP, Cr) or ions (Na) induced by ischemic injury be identified with novel, non-invasive imaging techniques?

CONTACTS AND LOCATIONS:
Overall Officials: Robert G. Weiss, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keceli G, Gupta A, Sourdon J, Gabr R, Schar M, Dey S, Tocchetti CG, Stuber A, Agrimi J, Zhang Y, Leppo M, Steenbergen C, Lai S, Yanek LR, O'Rourke B, Gerstenblith G, Bottomley PA, Wang Y, Paolocci N, Weiss RG. Mitochondrial Creatine Kinase Attenuates Pathologic Remodeling in Heart Failure. Circ Res. 2022 Mar 4;130(5):741-759. doi: 10.1161/CIRCRESAHA.121.319648. Epub 2022 Feb 3. PMID 35109669
- [Derived] Solaiyappan M, Weiss RG, Bottomley PA. Neural-network classification of cardiac disease from 31P cardiovascular magnetic resonance spectroscopy measures of creatine kinase energy metabolism. J Cardiovasc Magn Reson. 2019 Aug 12;21(1):49. doi: 10.1186/s12968-019-0560-5. PMID 31401975
- [Derived] Gabr RE, El-Sharkawy AM, Schar M, Panjrath GS, Gerstenblith G, Weiss RG, Bottomley PA. Cardiac work is related to creatine kinase energy supply in human heart failure: a cardiovascular magnetic resonance spectroscopy study. J Cardiovasc Magn Reson. 2018 Dec 10;20(1):81. doi: 10.1186/s12968-018-0491-6. PMID 30526611